CLINICAL TRIAL: NCT07074912
Title: Prescription Antipyretics to Decrease Unscheduled Return Visits In A Pediatric Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lina Palomares, Project Manager, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00006258
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Fever
Keywords: emergency department; fever; pediatrics
MeSH Terms: conditions — Fever; Emergencies | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescription for weight-based dosing of antipyretic (Experimental): The intervention group (n=220) will receive prescription with weight-based dosing for acetaminophen (also known and prescribed as Tylenol) and ibuprofen (also known and prescribed as Motrin).
  Interventions: Other: Prescription for weight-based dosing of antipyretic
- Standard discharge instructions (Active Comparator): The control group (n=220) will also receive standardized printed discharge instructions, which includes the appropriate dose of acetaminophen (also known as Tylenol) and ibuprofen (also known as Motrin) but no prescription.
  Interventions: Other: Standard discharge instructions

INTERVENTIONS:
Other: Prescription for weight-based dosing of antipyretic — The intervention group (n=220) will receive prescription with weight-based dosing for acetaminophen (also prescribed and known as Tylenol) and ibuprofen (also prescribed and known as Motrin).
  Arms: Prescription for weight-based dosing of antipyretic
Other: Standard discharge instructions — The control group (n=220) will also receive standardized printed discharge instructions but no prescription. The discharge instructions include the appropriate dose of acetaminophen (also known as Tylenol) and ibuprofen (also known as Motrin).
  Arms: Standard discharge instructions

SUMMARY:
The study aims to evaluate whether unscheduled return visits within one week for similar complaints are impacted by ensuring parents leave the emergency department (ED) with a prescription for appropriately dosed acetaminophen and ibuprofen for their child.

DETAILED DESCRIPTION:
Unscheduled return visits (URV) to the Emergency Department (ED) are a burden on both the healthcare system and patients. Published literature has attempted to categorize the rate of URV and type of complaints that lead to URVs. Rate of URV is variable, but as high as 22% for children with infectious illnesses and parents often return to the ED due to unresolved fever in a child. Unresolved fever may be due to continued progressive worsening of illness or inability to provide the appropriate amount of anti-pyretic (anti fever) medicine to the child, as pediatric medication dosing is not only age-based, but also weight-based. This increased variability could lead to confusion on the part of the caregivers. There are no published studies looking at whether appropriately prescribed antipyretics decrease the rate of return visits. Further, there is no standardization for antipyretic prescribing nationally or at the research team's hospital and some providers frequently provide prescriptions for these medications while others almost never do. It is unknown if providing a prescription for an over-the-counter medication makes a difference with health outcomes. The study aims to evaluate whether unscheduled return visits within one week for similar complaints are impacted by ensuring parents leave the ED with a prescription for appropriately dosed acetaminophen and ibuprofen.

This study will be a single center, randomized controlled trial in the pediatric emergency department (ED) at the north or central campus of Dell Children's Medical Center (DCMC). Patients meeting inclusion and exclusion criteria will be identified by research personnel during the ED visit.

Patients will be randomized to the intervention or control group after parental/caregiver permission is obtained for general participation in a research study. Computerized randomization functions and opaque envelopes will be used to achieve random assignment and allocation concealment. Patient care will look the same for all participants, but discharge process will differ slightly for each group. Both groups will receive standard discharge education, but the intervention group (n=220) will receive prescription with weight-based dosing for acetaminophen and ibuprofen. The control group (n=220) will also receive standardized printed discharge instructions, which includes the appropriate dose of acetaminophen and ibuprofen. As noted above, there is no standardization for antipyretic prescribing nationally or at our hospital. Some providers frequently provide prescriptions for these medications while others almost never do. It is unknown if providing a prescription for an over-the-counter medication makes a difference with patient satisfaction or health outcomes justifying the additional costs to the healthcare system.

One week after discharge, research personnel will contact participants to determine if an unscheduled return visit was made, and, if so, the reason why. Research personnel will ask about visits to EDs, urgent cares, and clinics/primary care providers, and about participant satisfaction with the care they received in the ED. The primary outcome will be unscheduled revisits to the ED (binary endpoint). Secondary endpoints include total number of unscheduled return visits, return with hospital admission, and parental satisfaction with ED care. The participant/caregiver will be debriefed on the randomization part of the study at this time and permission will be requested for continued use their child's health data and the caregiver's responses for the purposes of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to < 36 months of age being discharged home from Dell Children's Medical Center emergency department who are evaluated for fever
* Caregiver fluent in English or Spanish

Exclusion Criteria:

* Previous enrollment in this study
* Patient admitted to hospital
* Parental request for a prescription for acetaminophen and/or ibuprofen
* Trauma patient
* Orthopedic complaint
* Other painful indication for acetaminophen or ibuprofen
* Acetaminophen or ibuprofen prescribed for anything other than fever
* Allergy or another contraindication to acetaminophen or ibuprofen
* Parent and patient unlikely to follow up in the region (i.e., lives out of state)

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Unscheduled return visits | 7 days
  The primary outcome will be unscheduled revisits to the emergency department or urgent care (binary endpoint, i.e., yes/no). This information will be obtained directly from the caregiver/parent of the child. One week (7 days) after the initial visit to the emergency department, research personnel will call the parent/caregiver to ask about length of symptoms and any unscheduled return visits to the emergency department or urgent care for the same symptoms. Any return visits to an emergency department or urgent care will be noted as yes. Well child visits will not be counted.

SECONDARY OUTCOMES:
Parental satisfaction | 7 days
  Parental satisfaction with care received in the emergency department. Parents/caregivers will be contacted one week (7 days) after the initial visit to the emergency department and asked about their satisfaction with the visit ("How satisfied were you with the care your child received at the Dell Children's Medical Center Emergency Department?"). Responses are captured on a Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied) and parents/caregivers will be given an opportunity to expand on the level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wilkinson, MD, MPH, Study Director — The University of Texas at Austin
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared to protect patient confidentiality.

REFERENCES:
- [Background] Section on Clinical Pharmacology and Therapeutics; Committee on Drugs; Sullivan JE, Farrar HC. Fever and antipyretic use in children. Pediatrics. 2011 Mar;127(3):580-7. doi: 10.1542/peds.2010-3852. Epub 2011 Feb 28. PMID 21357332
- [Background] Trapani S, Fiordelisi A, Stinco M, Resti M. Update on Fever of Unknown Origin in Children: Focus on Etiologies and Clinical Approach. Children (Basel). 2023 Dec 24;11(1):20. doi: 10.3390/children11010020. PMID 38255334

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT07074912/Prot_SAP_000.pdf